CLINICAL TRIAL: NCT04384341
Title: Haemophilia and Bone Loss PHILEOS Study
Brief Title: Haemophilia and Bone Loss - PHILEOS Study
Acronym: PHILEOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 19PH224; 2019-A03358-49 (Other: ANSM)
Record Dates: First submitted 2020-05-05; First posted 2020-05-12 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Hemophilia
Keywords: Osteoporosis; fVIII; fIX; thrombin; Haemophilia; Hemophilia
MeSH Terms: conditions — Hemophilia A; Osteoporosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Haemophilic patients (Experimental): Blood sampling Bone Densitometry (BMD)
  Interventions: Radiation: Bone densitometry (BMD); Biological: Blood sampling for patients only
- Healthy volunteers (Other): Bone Densitometry (BMD)
  Interventions: Radiation: Bone densitometry (BMD)

INTERVENTIONS:
Radiation: Bone densitometry (BMD) — Recruitment of haemophilic patients during a routine visit at the haemophilia centre.
  Information of the subjects that the study requires a BMD measure for all and a blood sampling for patients only.
  After inclusion and exclusion criteria have been checked, the subject can sign the consent.
  For all subjects, an appointment will be made for BMD measure.
  For patients and controls: BMD will be measured by Dual Energy X-ray Absorptiometry (DXA) technology, on femoral and lumbar spine (L2-L4) sites.
  Recruitment of healthy volunteers through registers (Clinical Investigation Centers) and advertisements.
Biological: Blood sampling for patients only — For patients, fVIII/fIX activity and antigen, thrombin generation potential and plasmatic markers of bone remodelling will be measured centrally.
  Arms: Haemophilic patients

SUMMARY:
Haemophilia is a rare bleeding disorder, characterized by factor VIII (HA) or factor IX (HB) deficiency. The absence or the reduction of fVIII or fIX result in impaired thrombin generation and clot formation, causing excessive bleeding (mainly haemarthrosis). Osteoporosis is a systemic bone disease characterized by a low bone mineral density (BMD). A decrease of mean BMD has been described in haemophilic patients compared to healthy controls in several studies. So, osteoporosis could be an underestimated haemophilia-related comorbidity. None of the following risk factors (reduced physical activity, joint damage, vitamin D deficiency and /or hepatitis C virus (HCV) infection) has been retained as a cause of osteoporosis in haemophilic patients. Another hypothesis is that bone loss could be directly linked to fVIII or fIX and/or thrombin deficiency. The aim of this study is to evaluate the prevalence of the bone loss in HA and B patients, according to the type, the severity and the presence (or not) of a prophylactic treatment (depending on the age at which it was began) and to compare it to a control population. The investigators will also evaluate the relation between BMD and FVIII, fIX and thrombin potential.

DETAILED DESCRIPTION:
Recruitment of healthy volunteers through registers (Clinical Investigation Centers) and advertisements.

Recruitment of haemophilic patients during a routine visit at the haemophilia centre.

Information of the subjects that the study requires a BMD measure for all and a blood sampling for patients only.

After inclusion and exclusion criteria have been checked, the subject can sign the consent.

For all subjects, an appointment will be made for BMD measure. For patients and controls: BMD will be measured by Dual Energy X-ray Absorptiometry (DXA) technology, on femoral and lumbar spine (L2-L4) sites.

For patients, fVIII/fIX activity and antigen, thrombin generation potential and plasmatic markers of bone remodelling will be measured centrally.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers :

  * Healthy men aged between 20 to 60 years old
* Haemophilic Patients:

  * Haemophilia A and B patients, irrespective of the disease form (mild, moderate, severe with or without prophylaxis)
  * Haemophilic patients aged between 20 to 60 years old
  * Severe Haemophilia A patients with prophylaxis : last factor VIII injection more than 48 to 120 hours (depending on on the prophylactic treatment) prior blood sampling dedicated to the this research
  * Severe Haemophilia B patients : last factor IX injection more than 5 to 21 days (depending on the prophylactic treatment) prior blood sampling dedicated to the this research

Exclusion Criteria:

* Healthy Volunteers:

  * History of disease known to influence bone metabolism (hyperthyroidism, hyperparathyroidism, hypercorticism, hypogonadism, diseases that require long-term use of corticoids, …)
  * Past or present treatment with any osteoporotic medication other than Vit D or Ca++
  * Presence of two total hip prostheses
  * HIV documented infection
  * HCV documented infection (in progress or cured) at cirrhotic stage
* Haemophilic Patients:

  * Haemophilic patients with current or history of inhibitor anti-fVIII or anti-fIX (>5 Bethesda Units)
  * Treatment with HEMLIBRA (Emicizumab). Unless it is possible to use a result of thrombin generation prior to this treatment and achieved with a residual rate not greater than or equal to 5%.
  * History of disease known to influence bone metabolism and not related to haemophilia (hyperthyroidism, hyperparathyroidism, hypercorticism, hypogonadism, diseases that require long-term use of corticoids, …)
  * Past or present treatment with any anti-osteoporotic medication other than Vit D or Ca++
  * Presence of two total hip prostheses
  * HIV documented infection
  * HCV documented infection (in progress or cured) at cirrhotic stage

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 480 (Estimated)
Dates: Start 2020-06-02 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Osteoporosis defined by a T-score < -2.5 in severe haemophilic patients without prophylaxis and in healthy subjects. | During the procedure
  Bone mineral densitometry

SECONDARY OUTCOMES:
Osteoporosis defined by a T-score < -2.5 in the different groups of haemophilic patients and in in healthy subjects. | During the procedure
  Bone mineral densitometry
Osteopenia defined by a T-score < -1 in the different groups of haemophilic patients and in in healthy subjects. | During the procedure
  Bone mineral densitometry
Bone mineral density (expressed as a T-score) in the different groups of haemophilic patients and in healthy subjects. | During the procedure
  Bone mineral densitometry
Basal level of fVIII/fIX (expressed as an Ag level or as a %) or thrombin generation potential (expressed as an endogenous thrombin potential (ETP), nmol/min) and Bone mineral density (expressed as a T-score and Z-score) | At the inclusion
  Blood test Relation between the basal level of fVIII or fIX (expressed as an Ag level or as a %) or the thrombin generation potential (expressed as an endogenous thrombin potential (ETP), nmol/min) and Bone mineral density (expressed as a T-score and Z-score)
Markers influencing bone metabolism in all haemophilic patients included | At the inclusion
  Blood test

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte TARDY, MD, Principal Investigator — CHU de Saint Etienne
Locations (23):
- BELGIUM - Brussels, Brussels, Belgium
- University Hospital Centre Zagreb, Zagreb, Croatia
- France (19):
  - Chu de Bordeaux, Bordeaux
  - Chu Brest Hopital Morvan, Brest
  - HCL - Groupement Hospitalier Est (Hôpital Louis Pradel), Bron
  - CHU Caen, Caen
  - Centre Hospitalier Metropole Savoie, Chambéry
  - Chu Cth Estaing Clermont Ferrand, Clermont-Ferrand
  - Chu de Dijon, Dijon
  - Chu Grenoble Alpes, Grenoble
  - CHU Lille, Lille
  - Chu La Timone Marseille, Marseille
  - CHU - Saint Eloi, Montpellier
  - CHU Nancy, Nancy
  - CHU de Nantes, Nantes
  - Chu Necker Paris, Paris
  - APHP - Bicêtre, Paris
  - Chu Rennes Hopital Pontchaillou, Rennes
  - CHU de ROUEN, Rouen
  - CHU de Saint-Etienne, Saint-Etienne
  - Chu Strasbourg - Hôpital de Hautepierre, Strasbourg
- MHEK, Budapest, Hungary
- ROMANIA - Bucharest, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tardy-Poncet B, Play B, Montmartin A, Damien P, Ollier E, Presles E, Garcin A, Tardy B. PHILEOS (haemoPHILia and ostEoporOSis) Study: protocol of a multicentre prospective case-control study. BMJ Open. 2021 Jan 13;11(1):e042283. doi: 10.1136/bmjopen-2020-042283. PMID 33441362